CLINICAL TRIAL: NCT02514265
Title: MAPP Research Network: Trans-MAPP Study of Urologic Chronic Pelvic Pain: Symptom Patterns Study (SPS)
Brief Title: Trans-MAPP Symptom Patterns Study (SPS)
Acronym: MAPP II SPS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 822352; 5U01DK082316-02 (NIH)
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Interstitial Cystitis; Chronic Prostatitis
Keywords: pelvic pain, bladder pain
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA Blood Urine Vaginal Swabs Rectal Swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UCPPS patients: All participants in this study are men or women who have been diagnosed with Urologic Chronic Pelvic Pain Syndrome (UCPPS). Approximately one-half of the participants will be male, and one-half will be enriched to meet the body map pain location criteria of pelvic pain (PP) only. In addition, enrichment recruitment of 240 UCPPS patients (120 males; 120 females) will also be targeted for those who answer "no" to questionaire question about specific Bladder pain symptoms.

SUMMARY:
This study is the second phase of the MAPP Network and is designed to conduct a prospective, observational study of men and women with UCPPS, referred to as the Symptom Patterns Study (SPS), enriched with pre-defined subgroups, with longer follow-up, in order to further investigate clinical and biologic factors associated with worsening and/or improvement of reported urinary and non-urinary symptoms.

DETAILED DESCRIPTION:
To better understand the etiology and treated natural history of UCPPS, and to identify clinical factors and research measurements to define clinically relevant sub-groups of these patients for future clinical trials, and to inform symptom management, the NIDDK established the Multidisciplinary Approach to the Study of Chronic Pelvic Pain (MAPP) Research Network in 20089 (http://www.mappnetwork.org/). The primary clinical research effort carried out by this network in Phase I was a prospective cohort study, the Trans-MAPP Epidemiology/Phenotyping (EP) Study.10 From 12/14/2009 through 12/14/2012 1,039 men and women were enrolled, including persons with UCPPS (n=424); persons with other co-morbid illnesses, including fibromyalgia, irritable bowel syndrome, and chronic fatigue syndrome (n=200 for all conditions); and healthy controls (n=415). Study participants were extensively characterized (i.e., phenotyped) at baseline, and UCPPS participants were followed for 12 months. During follow-up, using a web-based symptom data capture system, a small battery of self-report questionnaires were repeated on a bi-weekly schedule for 48 weeks. In addition, neuroimaging was performed in a subset of participants (n=279) at baseline, and biological samples were collected on all participants at baseline and follow-up for studies to identify plasma and urine biomarkers and potential infectious agents. This study was complemented by a number of Discovery Site-Specific clinical research studies (i.e., studies generally conducted at a single site) and investigations of animal models developed by multiple sites to mimic symptoms of human UCPPS.

Initial analyses of these data have identified a number of provocative findings. There are strong indications those certain subgroups of participants (albeit with small sample sizes) with urinary and non-urinary symptoms tend to improve over time; whereas other subgroups tend to worsen over time. These patterns of improving or worsening are differentially expressed according to sex, subtype of bladder pain syndrome (BPS), and pain location (localized to the pelvic region vs pain reported in the pelvic region and beyond).

The second phase of the MAPP Network is designed to conduct a prospective, observational study of men and women with UCPPS, referred to as the Symptom Patterns Study (SPS). This follow-up study will have pre-defined subgroups, with longer follow-up, in order to further investigate clinical and biologic factors associated with worsening and/or improvement of reported urinary and non-urinary symptoms.

This proposed MAPP Phase II SPS also presents the opportunity to apply many of the most promising research methods in the pain field (e.g. functional, chemical and structural neuroimaging, quantitative sensory testing) during the course of the study (at baseline and then longitudinally) to better characterize men and women with UCPPS. Most of these measures were only collected at a single point in time in the Trans-MAPP Epidemiology/Phenotyping Study of Phase I, and within a sample of UCPPS patients not enriched with predefined subgroups. Further phenotyping in the second phase study will allow us to better determine which of these measures, or any other measures identified during Phase I (e.g., urinary or serum biomarkers), might identify individuals most likely to have spontaneous improvement of their symptoms, versus transition to a more "peripheral" (pelvic pain only) or "centralized" form (pelvic pain and beyond) of urinary and non-urinary pain.

Eligible participants will be asked to participate in the study for up to 36 months. During which they will be asked to complete a series of in-clinic study visits that will at various time points a neuroimaging scan and quantitative sensory tests, online internet-based questionnaires in clinic and off site/at home (assessing symptoms, health care utilization, flare status, and quality of life), a physical exam, a pelvic exam, and prostate massage (optional for males only).

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for the SPS if they meet the following criteria:

1. Participant has signed and dated the appropriate Informed Consent document.

   * Agreed to participate in ALL required Symptoms Patterns Study procedures (including Biospecimen collections, Neuroimaging, and Quantitative Sensory Testing).
   * Gave permission for use of DNA for genetics studies.
2. Participant is at least 18 years of age.
3. Participant is able to speak, read, and understand English.
4. In the past 3 months participant has had a feeling of pain, pressure, or discomfort in the lower abdomen or pelvic area -- that is, the part of the body that is above the participant's legs and below the belly button.
5. These symptoms have been present for the majority of the time during the most recent 3 months.
6. Participant reports a response of at least 1 on the pain, pressure or discomfort scale for UCPPS symptoms during the past 2 weeks.
7. Participant has received a clinical diagnosis of either or both IC/BPS or CP/CPPS (per AUA guidelines) or a clinician familiar with UCPPS criteria confirms participant meets UCPPS evaluation criteria per-protocol.

Exclusion Criteria:

Any patient meeting any one of the following criteria will not be eligible for enrollment in the Symptom Patterns Study. However, participants who develop any of these exclusion criteria during the follow-up phase of the study will continue to be followed. It will be recorded in the follow-up data if a patient has developed any of the exclusion criteria.

1. Participant has an on-going symptomatic urethral stricture.
2. Participant has an on-going neurological disease or disorder affecting the bladder or bowel fistula.
3. Participant has a history of cystitis caused by tuberculosis, radiation therapy or Cytoxan/cyclophosphamide therapy.
4. Participant has augmentation cystoplasty or cystectomy.
5. Participant has an active autoimmune or infectious disorder (such as Crohn's Disease or Ulcerative Colitis, Lupus, Rheumatoid Arthritis, Multiple Sclerosis, or HIV).
6. Participant has a history of cancer (with the exception of skin cancer).
7. Participant has current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc.).
8. Participant has severe cardiac, pulmonary, renal, or hepatic disease that in the judgment of the study physician would preclude participation in this study.

Exclusion Criteria for Males Only

1. Diagnosis of unilateral orchalgia, without pelvic symptoms.
2. History of transurethral microwave thermotherapy (TUMT), transurethral needle ablation (TUNA), balloon dilation, prostate cryo-surgery, or laser procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Trans-MAPP SPS study will include adults 18 years and older with urological pelvic pain syndromes. Approximately one-half of the participants will be male, and one-half will be enriched to meet the body map pain location criteria of Pelvis pain only.
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Pain Severity Score | 48 weeks
  The Pain severity Score is constructed from the GUPI pain subscale score (0-23) and ICSI Q4: Bladder pain score (0-5), summed to create a primary outcome for UCPPS pain, ranging from 0 to 28.
Urinary Severity Score | 48 weeks
  The Urinary Severity Score is constructed from the GUPI urinary subscale score (0-10) and sum of ICSI Q1: Strong need to urinate (0-5), ICSI Q2: Frequency (0-5), and ICSI Q3: Frequency at night (0-5), summed to create a primary outcome for urinary symptoms, ranging from 0 to 25.

CONTACTS AND LOCATIONS:
Overall Officials: J.Quentin Clemens, MD, MSCI, Study Chair — University of Michigan; Chris Mullins, PhD, Study Director — NIDDK, NIH; J. Richard Landis, PhD, Study Director — University of Pennsylvania, DCC
Locations (6):
- United States (6):
  - University of California Los Angeles/University of Southern California, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St. Louis, St Louis, Missouri
  - University of Washington, Seattle, Seattle, Washington

REFERENCES:
- [Derived] Schrepf A, Locke K, Moldwin R, Williams DA, Till S, Farrar J, Richard Landis J, Tu F, Rodriguez L, Lai H, Naliboff B, Kutch J, Harte SE, Harris RE, Kreder KJ, Spitznagle T, McKernan L, Yang C, Quentin Clemens J, Mullins C, Clauw DJ. Widespread Pain Moderates the Response to Centrally-Acting Therapies in an Observational Cohort of Patients With Urologic Chronic Pelvic Pain Syndrome: A MAPP Research Network Study. Neurourol Urodyn. 2025 Aug;44(6):1290-1295. doi: 10.1002/nau.70068. Epub 2025 May 25. PMID 40415481
- [Derived] Naliboff BD, McWilliams T, Clemens JQ, Pontari MA, Stephens-Shields AJ, Moldwin R, Sutcliffe S, Mullins C, Landis JR. Relationship of Sex and Diagnosis With Symptoms and Illness Impact in Urologic Chronic Pelvic Pain; A Mapp Network Analysis. Neurourol Urodyn. 2025 Feb;44(2):400-408. doi: 10.1002/nau.25648. Epub 2024 Dec 20. PMID 39704257
- [Derived] Leech KA, Kettlety SA, Mack WJ, Kreder KJ, Schrepf A, Kutch JJ. Brain predicted age in chronic pelvic pain: a study by the Multidisciplinary Approach to the Study of Chronic Pelvic Pain Research Network. Pain. 2025 May 1;166(5):1060-1069. doi: 10.1097/j.pain.0000000000003424. Epub 2024 Oct 16. PMID 39432808
- [Derived] Schrepf AD, Mawla I, Naliboff BD, Gallop B, Moldwin RM, Tu F, Gupta P, Harte S, Krieger JN, Yang C, Bradley C, Rodriguez L, Williams D, Magnotta V, Ichesco E, Harris RE, Clemens Q, Mullins C, Kutch JJ. Neurobiology and long-term impact of bladder-filling pain in humans: a Multidisciplinary Approach to the Study of Chronic Pelvic Pain (MAPP) research network study. Pain. 2023 Oct 1;164(10):2343-2351. doi: 10.1097/j.pain.0000000000002944. Epub 2023 Jun 6. PMID 37278657
- [Derived] Schrepf A, Kaplan C, Harris RE, Williams DA, Clauw DJ, As-Sanie S, Till S, Clemens JQ, Rodriguez LV, Van Bokhoven A, Landis R, Gallop R, Bradley C, Naliboff B, Pontari M, O'Donnell M, Luo Y, Kreder K, Lutgendorf SK, Harte SE. Stimulated whole-blood cytokine/chemokine responses are associated with interstitial cystitis/bladder pain syndrome phenotypes and features of nociplastic pain: a multidisciplinary approach to the study of chronic pelvic pain research network study. Pain. 2023 May 1;164(5):1148-1157. doi: 10.1097/j.pain.0000000000002813. PMID 36279178
- [Derived] Naliboff BD, Schrepf AD, Stephens-Shields AJ, Clemens JQ, Pontari MA, Labus J, Taple BJ, Rodriguez LV, Strachan E, Griffith JW. Temporal Relationships between Pain, Mood and Urinary Symptoms in Urological Chronic Pelvic Pain Syndrome: A MAPP Network Study. J Urol. 2021 Jun;205(6):1698-1703. doi: 10.1097/JU.0000000000001595. Epub 2021 Feb 4. PMID 33535797
- See also: MAPP Research Network Website — http://www.mappnetwork.org/